CLINICAL TRIAL: NCT05598268
Title: A Phase I/IIa Study to Assess the Safety, Tolerability, Biodistribution and Pharmacodynamic of T3011 Herpes Virus Administered Via Intravenously in Patients With Advanced Solid Tumors.
Brief Title: A Study of T3011 Administered Via Intravenously in Patients With Advanced Solid Tumors.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmVira Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MVR-T3011-002
Record Dates: First submitted 2022-10-18; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumor; Lung Cancer; Liver Cancer; Lymphoma; Mesothelioma of Pleura
Keywords: Herpes virus; Advanced solid tumor; Dose escalation; T3011; Oncolytic virus
MeSH Terms: conditions — Lung Neoplasms; Liver Neoplasms; Lymphoma; Mesothelioma, Malignant

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T3011 Herpes Virus Injection (Experimental)
  Interventions: Biological: T3011

INTERVENTIONS:
Biological: T3011 — T3011 will be administered through IV drip

SUMMARY:
This is a multicenter, open-label study conducted in 3 phases:

Dose escalation stage: The stage contain 4 cohorts, each cohort divided into 2 groups （group A, single dose and Group B, multiple dose）.Dose escalation will use a 3+3 design to evaluate escalating doses of T3011.Cohorts of three subjects will be enrolled at each T3011 dose level with expansion to six subjects, if necessary, to assess toxicity. Total enrollment will depend on the toxicities observed, with approximately 4-24 evaluable subjects enrolled in dose escalation stage.

Dose extension stage: The SMC will evaluate the available safety and preliminary efficacy data and initiate dose-expansion studies for the appropriate indications Phase IIa: To explore the safety of intravenous administration and expand the study in other indications. the stage will be carried out gradually based on the data obtained from the phase I study.

DETAILED DESCRIPTION:
This is a multicenter, open-label study conducted in 3 phases:

Dose escalation stage: The stage contains 4 cohorts, divided into cohort 1 (1x106PFU/ dose), cohort 2 (1x107PFU/ dose), cohort 3 (1x108PFU/ dose) and cohort 4 (3x108PFU/ dose). Each cohort divided into 2 groups （group A, single dose and Group B, multiple dose）.Dose escalation will use a 3+3 design to evaluate escalating doses of T3011. At any dose level, if no DLT occurs among the first 3 subjects, then escalation to the next dose level may proceed, with the approval of the SMC. If 1 DLT occurs in the first 1 to 3 subjects, the dose level will expand to a maximum of 6 subjects. If no DLT occurs among the additional subjects, then escalation to the next dose level may proceed, with the approval of the SMC. If 2 or more DLTs occur within a cohort, then that dose level will be above the maximum tolerated dose (MTD) (the highest dose where no more than 1 of 6 subjects has experienced a DLT), and new subjects will be enrolled at the previous lower (tolerated) dose level until that cohort has 6 subjects. This lower dose level will be considered the MTD if ≤ 1 in 6 subjects has a DLT. At the end of dose escalation, the SMC will recommend a dose (the recommended phase 2 dose [RP2D]) of T3011 to be used in phase 2a expansion study based upon MTD identification, cumulative safety, pharmacokinetic (PK), efficacy, and pharmacodynamic data. Total enrollment will depend on the toxicities observed, with approximately 4-24 evaluable subjects enrolled in dose escalation stage.

In group A, participant will receive a single dose and the DLT evaluation period is 14 days.

In group B, Participants will receive administration at D1/D4/D8 of every cycle. The DLT evaluation period will be the first 21-day Cycle in group B. Tumor evaluation was performed every two cycles. The maximum treatment period should not exceed 4 cycles. Group B of cohort X was enrolled only after the DLT assessed for group A of cohort X and SMC approval to proceed to the next cohort assessment.

Dose extension stage: The SMC will evaluate the available safety and preliminary efficacy data and initiate dose-expansion studies for the appropriate indications Phase IIa: To explore the safety of intravenous administration and expand the study in other indications. the stage will be carried out gradually based on the data obtained from the phase I study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Locally recurrent or metastatic solid tumors, There is currently no effective treatment (including treatment intolerance).

  2. Age 18 years or older. 3. At least one target lesion per RECIST version 1.1. 4. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1. 5. Life expectancy ≥ 12 weeks. 6. Women of childbearing potential must have a negative serum pregnancy test at Screening within 7 days of dosing with T3011.

  7. Understand and sign ICF voluntarily,capable of understanding and complying with protocol requirements.

Exclusion Criteria:

* 1. Pregnant or lactating or plan to pregnant or give birth during the trial. 2. Splenectomy, previous allogenic organ transplant. 3. Prior treatment with another gene therapy（except T3011）. 4. Requires continued concurrent systemic therapy with any drug active against HSV (acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir). Topical use of drugs against HSV are allowed.

  5. History of allergic reactions attributed to compounds of similar biological composition to HSV-1, IL-12, or anti-PD-1 monoclonal antibody or their excipients.

  6. Prior treatment with anti-PD-(L)1 monoclonal antibody in combination with IL-12.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of escalating doses of IV T3011 in Patients with advanced malignant tumors | Up to 2 years from first dose of T3011
  Incidence of AE(TEAE)
Assess DLTs and identify the RP2D of single agent IV T3011 | Up to 2 years from first dose of T3011
  Incidence of DLT
Assess safety and tolerability of T3011 intravenous administration at MTD or RP2D doses through dose extension study | Up to 2 years from first dose of T3011
  Incidence of AE(TEAE)

SECONDARY OUTCOMES:
Evaluate the biodistribution and viral shedding of IV T3011 | Up to 2 years from first dose of T3011
  Measurement of T3011 in subjects' blood, urine, and saliva for biodistribution and viral shedding
Evaluate the immunogenicity of IV T3011 | Up to 2 years from first dose of T3011
  Measurement of ADAs and Nabs of IL-12, anti-PD-1 antibody and HSV-1 (test Nabs when ADAs are positive).
Evaluate the preliminary clinical response of single agent IV T3011 | Up to 2 years from first dose of T3011
  ORR PFS and OS

OTHER OUTCOMES:
Exploring tumor immunomodulatory mechanism | Up to 42 days from first dose of T3011
  Lymphocyte typing
Exploring histological changes after IT T3011 | Up to 42 days from first dose of T3011
  Immunofluorescence detection
Exploring the relationship between genetic changes and drug efficacy | Up to 42 days from first dose of T3011
  Tumor tissue sequencing

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital of Bengbu Medicial College, Bengbu, Anhui
  - Zhujiang Hospital of Southern Medical University, Guanzhou, Guangdong
  - the First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hosptial, Zhengzhou, Henan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Beijing Chest Hospital, Beijing
  - Shanghai Chest Hosptial, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided